CLINICAL TRIAL: NCT00105469
Title: A Study to Evaluate the Clinical and Microbial Efficacy and Safety of 1.0% AzaSite Compared to 0.3% Tobramycin Ophthalmic Solution in the Treatment of Bacterial Conjunctivitis
Brief Title: Evaluation of Clinical and Microbial Efficacy and Safety of AzaSite Compared to Tobramycin for Bacterial Conjunctivitis (C-01-401-004)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Vice President, Late Stage Development Group Leader, Merck Sharp & Dohme Corp
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P08633; C-01-401-004
Record Dates: First submitted 2005-03-14; First posted 2005-03-15 (Estimated); Results first posted 2011-10-27 (Estimated); Last update posted 2013-12-16 (Estimated); Status verified 2013-11

CONDITIONS: Bacterial Conjunctivitis
Keywords: Bacterial Conjunctivitis; Pink Eye; Conjunctivitis; Eye Infection
MeSH Terms: conditions — Conjunctivitis, Bacterial; Conjunctivitis; Eye Infections | interventions — Azithromycin; Tobramycin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- AzaSite (Experimental): 1.0% azithromycin in DuraSite
  Interventions: Drug: AzaSite
- Tobramycin (Active Comparator): 0.3% tobramycin
  Interventions: Drug: Tobramycin

INTERVENTIONS:
Drug: AzaSite — AzaSite ophthalmic solution; one topical drop to the infected eye or eyes twice daily (in the morning and at bedtime) on Days 1 and 2 followed by once daily (in the morning between 7 and 10am) on Days 3 through 5.
  Arms: AzaSite
Drug: Tobramycin — Tobramycin ophthalmic solution; one topical drop to the infected eye or eyes four times daily at 4 to 6 hour intervals (first dose in the morning between 7 and 10am) for 5 days.
  Arms: Tobramycin

SUMMARY:
The purpose of this study is to evaluate the clinical and microbial efficacy and safety of AzaSite compared to tobramycin for bacterial conjunctivitis. Adults and children one year of age and older with bacterial conjunctivitis in at least one eye are eligible. Subjects will be randomly assigned to the AzaSite group or Tobramycin group. Three visits will be required for the study.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subject, of any race, who is at least 1 year of age.
* Subjects must have a clinical diagnosis of acute bacterial conjunctivitis and exhibit mucopurulent or purulent conjunctival discharge (crusty or sticky eyelids, globular and yellow discharge) and redness in at least one eye.
* The symptoms of bacterial conjunctivitis must be present for 3 days (approximately 72 hours) or less.
* Must be willing to discontinue contact lens wear for the duration of the study.

Exclusion Criteria:

* Any uncontrolled systemic disease or debilitating disease.
* Use of topical ophthalmic solutions including tear substitutes within 2 hours before and during the study.
* Use of any topical ophthalmic anti-inflammatory agents within 48 hours before and during study.
* Any active upper respiratory tract infection.
* Pregnant or nursing females.
* Use of any antibiotic (topical or systemic) within 72 hours of enrollment.

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 743 (Actual)
Dates: Start 2004-07; Primary Completion 2005-10 (Actual); Study Completion 2005-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (26):
- United States (26):
  - Renaissance Center, Birmingham, Alabama
  - Children's Eye Physicians, Littleton, Colorado
  - Palm Beach Eye Associates, Atlantis, Florida
  - The Eye Associates, Bradenton, Florida
  - Alan Shuster, MD, Jupiter, Florida
  - Pasco Eye Institute, New Port Richey, Florida
  - Tukoi Institute for Clinical Research, North Miami Beach, Florida
  - Advanced Eye Care, Panama City, Florida
  - Presidential Eye Center, West Palm Beach, Florida
  - Jon Fishburn, MD, Boise, Idaho
  - Medisphere Medical Research Center, LLC, Evansville, Indiana
  - Hutchinson Clinic, Hutchinson, Kansas
  - Massachusetts Eye and Ear Infirmary, Boston, Massachusetts
  - Mason Eye Institute, Columbia, Missouri
  - Ophthalmology Associates, Creve Coeur, Missouri
  - Research Eye Care Center, Kansas City, Missouri
  - Ophthalmology Associates, Princeton, New Jersey
  - Huntington Medical Group, Huntington Station, New York
  - Cornerstone Eye Care, High Point, North Carolina
  - Eye Health Northwest, Portland, Oregon
  - Irving Weinberger, MD, Pittsburgh, Pennsylvania
  - Southern Eye Associates, PA, Greenville, South Carolina
  - Corona Research Consultants, Inc., El Paso, Texas
  - Cottonwood Ophthalmology Associates, Murray, Utah
  - Rockwood Clinic, PS-Eye Center, Spokane, Washington
  - Wenatchee Valley Medical Center, Wenatchee, Washington

REFERENCES:
- [Derived] Protzko E, Bowman L, Abelson M, Shapiro A; AzaSite Clinical Study Group. Phase 3 safety comparisons for 1.0% azithromycin in polymeric mucoadhesive eye drops versus 0.3% tobramycin eye drops for bacterial conjunctivitis. Invest Ophthalmol Vis Sci. 2007 Aug;48(8):3425-9. doi: 10.1167/iovs.06-1413. PMID 17652708
- See also: Related Info — http://www.insitevision.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | AzaSite | Tobramycin
Started | 365 | 378
Completed | 343 | 367
Not Completed | 22 | 11
Not completed — Adverse Event | 9 | 8
Not completed — Protocol Violation | 4 | 0
Not completed — Withdrawal by Subject | 2 | 3
Not completed — Lost to Follow-up | 1 | 0
Not completed — Lack of Efficacy | 2 | 0
Not completed — Other Reason | 4 | 0

BASELINE CHARACTERISTICS:
Groups:
- AzaSite; Tobramycin: Per protocol population (defined as all randomized
  subjects who had administered at least one drop of the appropriate study drug, demonstrated evidence of
  pathogenic bacteria levels, presented clinical signs of conjunctivitis at Visit 1, and returned for at least one post-first dose clinical assessment) with last observation carried forward.
- Total: Total of all reporting groups
Arm/Group | AzaSite | Tobramycin | Total
Number analyzed (Participants) | 159 | 157 | 316
Age, Continuous [Mean (Standard Deviation); unit: years] | 17.9 (20.23) | 22.8 (22.61) | 20.4 (21.55)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 81 | 90 | 171
  Male | 78 | 67 | 145

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Achieved Clinical Resolution at Visit 3
Description: Clinical resolution is defined as absence of all three clinical signs (ocular discharge, bulbar conjunctival injection, and palpebral conjunctival injection).
Time Frame: Visit 3 (Day 6)
Population: Per protocol population (defined as all randomized
  subjects who had administered at least one drop of the appropriate study drug, demonstrated evidence of
  pathogenic bacteria levels, presented clinical signs of conjunctivitis at Visit 1, and returned for at least one post-first dose clinical assessment) with last observation carried forward.
Measure: Number; unit: Participants
Arm/Group | AzaSite | Tobramycin
Number analyzed (Participants) | 159 | 157
Participants | 127 | 123

2. Secondary Outcome: Number of Participants Who Achieved Bacterial Eradication at Visit 3
Description: Bacterial eradication is defined as eradication of the causative pathogens as indicated by the absence of growth (0 colony forming units/mL) of the original infecting organism(s).
Time Frame: Visit 3 (Day 6)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | AzaSite | Tobramycin
Number analyzed (Participants) | 159 | 157
Participants | 140 | 148

ADVERSE EVENTS:
Arm/Group | AzaSite | Tobramycin
Serious Adverse Events (participants affected / at risk) | 0/365 | 0/378
Other Adverse Events (participants affected / at risk) | 0/365 | 0/378

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institution and Principal Investigator shall not publish, present or use any data or results arising out of the performance of this study for their own instruction, research or publication without the prior express written consent of Sponsor.